CLINICAL TRIAL: NCT01345890
Title: Neuromodulation in Post Stroke Dysphagia
Brief Title: Cortical Neuromodulation in Post Stroke Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2004/008/HP
Record Dates: First submitted 2009-02-17; First posted 2011-05-02 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Dysphagia
Keywords: swallowing; stroke; aspiration; human; electrical stimulation; post stroke dysphagia
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- electrical stimulation (Experimental): stroke patients
  Interventions: Procedure: electrical stimulation

INTERVENTIONS:
Procedure: electrical stimulation — sub motor threshold stimulation of mylohyoid muscles

SUMMARY:
The investigators aim is to try to rehabilitate post stroke dysphagia using electrical stimulation of the mylohyoid muscles.

DETAILED DESCRIPTION:
Aspiration could have fatal complication especially in post stroke dysphagia. The aim of this study is to improve post stroke dysphagia using electrical stimulation of mylohyoid muscles.

The investigators measure swallowing time before and after electrical stimulation, performed one hour per day, 5 consecutive days during paste consistency swallowing

ELIGIBILITY:
Inclusion Criteria:

* post stroke dysphagia

Exclusion Criteria:

* contraindication to magnetic stimulation, unability to accept the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
videofluoroscopy | before and after (once a day for 5 consecutive days)
  measure swallowing time before and after electrical stimulation, performed one hour per day, 5 consecutive days during paste consistency swallowing

CONTACTS AND LOCATIONS:
Overall Officials: Eric VERIN, MD-PhD, Principal Investigator — Rouen University
Locations (1):
- Rouen Universty Hospital, Rouen, France